CLINICAL TRIAL: NCT05337683
Title: A Retrospective Non-Interventional Study to Evaluate the Impact of Eculizumab in Korean Paroxysmal Nocturnal Hemoglobinuria Patients
Brief Title: A Retrospective Non-Interventional Study to Evaluate the Impact of Eculizumab in Korean PNH Patients
Status: Completed | Type: Observational
Sponsor: Handok Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: HD_ECU_OS2020
Record Dates: First submitted 2022-04-08; First posted 2022-04-20 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: PNH

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a retrospective non-interventional study, and the main objective of this study is to identify the impact of eculizumab treatment and the improvement of complications before and after eculizumab treatment, and to evaluate the safety during the treatment and the clinical unmet needs during the treatment in PNH patients in real-world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with PNH aged 18 years or older who started eculizumab treatment in accordance with drug label between 2012 and January 31st, 2020. (However, patients who have received eculizumab as part of a clinical trial or an expanded access program/compassionate use program prior to 2012 are also eligible.)
* Patients who are vaccinated against Neisseria meningitidis at least 2 weeks prior to starting eculizumab treatment. Patients who have been treated with appropriate prophylactic antibiotic therapy for 2 weeks after vaccination if they received eculizumab within 2 weeks after the vaccination.

Exclusion Criteria:

* Pediatric patients with PNH aged under 18 years
* Patients with hypersensitivity to the active ingredients of eculizumab, murine protein, or other components
* Patients with untreated severe meningococcal (Neisseria meningitidis) infection
* Patients who received other complement inhibitors for PNH before or during eculizumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PNH aged 18 years or older who started receiving eculizumab treatment accordance with the drug label until January 31, 2020 will be enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-08-30 (Actual); Study Completion 2022-01-03 (Actual)

PRIMARY OUTCOMES:
Decrease of hemolysis after eculizumab treatment | The results of LDH tests performed before eculizumab treatment, at 6, 12, 24 months after the start of eculizumab treatment, and every 12 months thereafter will be collected.
  The change in LDH levels before and after eculizumab treatment will be compared to determine whether hemolysis decreased after the treatment.
The Improvement/occurrence of complications and related clinical symptoms before and after eculizumab treatment | 6 months before eculizumab administration to the end of the administration (It is up to subject's treatment period. Through study completion, an average of 51months)
  The major complications due to PNH include thromboembolism, pulmonary hypertension, renal failure, and smooth muscle spasm, and their occurrence will be determined by the investigator.
  In addition, PNH-related symptoms (fatigue, anemia, dysphagia, shortness of breath/dyspnea, chest pain, abdominal pain, erectile dysfunction, hemoglobinuria, others) before and after eculizumab administration will be compared.
Severity of anemia | Before the administration, at 6, 12, 24 months after the start of the treatment and every and 12 months thereafter
  Hb levels will be compared to identify the severity of anemia.
The required Unit of pRBC transfusion before and after eculizumab treatment | From 1 year before the treatment to the end of the administration (It is up to subject's treatment period. Through study completion, an average of 51months)
Effectiveness Evaluation at Last Follow-Up | At the last follow-up (At the time of data collection retrospectively)
  The investigator will perform the final evaluation of the efficacy for entire observation period based on the collected data. The investigator will comprehensively judge and evaluate the decrease of hemolysis occurrence, the improvement and occurrence of complications, and the severity of anemia, etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Handok, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No